CLINICAL TRIAL: NCT04173585
Title: TEAM-Trial: Targeting Epigenetic Therapy Resistance in AML With Bortezomib: A Multi-centre Matched Threshold Crossing Phase II Approach
Brief Title: TEAM-Trial: Targeting Epigenetic Therapy Resistance in AML With Bortezomib
Acronym: TEAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard F Schlenk, Scientific Coordinator, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2017-0530
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; therapy resistance; refractory/relapsed; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Bortezomib; Gemtuzumab

STUDY DESIGN:
Intervention Model Description: Simon's Optimal Two-Stage Design: The Matched Threshold Crossing (MTC) Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bortezomib-Gemtuzumab Ozogamicin Treatment (Experimental): one cycle of combined chemotherapy:
  * Bortezomib (1.3 mg/m2) sc on day 1 and 3. Dose will be given 3 hours prior to Cytarabine on day 1 and 3
  * Cytarabine (1g/m² twice daily) iv over 3 hours on day 1, 2 and 3 Gemtuzumab Ozogamicin (3 mg/m²,up to a maximum of one 5 mg vial) iv over 2 hours on day 1 after first dose of Cytarabine and day 4
  * Pegfilgrastim 6 mg sc on day 8 (optional)
  Interventions: Drug: Bortezomib; Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: Bortezomib — Bortezomib is a small molecule dipeptide binding the catalytic site of the 26 S proteasome. It acts as a potent, reversible, and specific inhibitor of proteasomes and thus impairs the degradation of ubiquitinated proteins. It has demonstrated anti-neoplastic activity in myeloma and lymphoma. It is approved and widely used in multiple myeloma both for first line treatment and relapsed patients.
  Other Names: Velcade
Drug: Gemtuzumab Ozogamicin — Gemtuzumab Ozogamicin is a monoclonal antibody directed against the myeloid surface antigen CD33. The antibody is linked to calicheamicin which serves as cytotoxic agent. For years, gemtuzumab ozogamicin has been tested in clinical AML trials. Though withdrawn from the US market in 2010, FDA approval was granted in September 2018, EU approval in April 2018 based on encouraging results from recent clinical trials using enhanced dosing schedules.
  Other Names: Mylotarg

SUMMARY:
The long-term outcome of patients with acute myeloid leukemia (AML) remains poor, with less than 30% of patients achieving long lasting remission or cure. This poor outcome is largely due to refractoriness to induction chemotherapy as well as relapses during and after completion of intensive induction and consolidation therapy. In patients with refractory/relapsed AML hematopoietic cell transplantation (allo-HCT) is currently the only treatment option offering a prospect of cure but outcome is heavy influenced by the remission status before allo-HCT. Therefore, patients are typically treated with salvage regimens based on high dose cytarabine (HiDAC) combined with mitoxantrone, fludarabine or idarubicin. Nevertheless, the remission rates remain poor and currently there is no accepted standard salvage regimen. Recent studies indicate that combination chemotherapy including HiDAC and gemtuzumab ozogamicin (GO) at a dose of 3 mg/m² leads to improved response rates in refractory AML.

Proteasome inhibition with bortezomib appears to be a promising treatment strategy to restore chemo-sensitivity via EZH2 stabilisation.

This study aims at improving response rates in refractory/ relapsed AML by combining high dose cytarabine, gemtuzumab ozogamicin (GA) and bortezomib (B).

During this phase II study efficacy of B-GA is assessed in comparison to matched historical controls using the Matched Threshold Crossing (MTC)-approach. If results are promising, a subsequent randomized phase III study is intended to assess the efficacy of GA with or without bortezomib.

DETAILED DESCRIPTION:
Acute Myeloid Leukemia (AML) is a clonal malignant disorder which is characterized by the expansion of leukemic blasts in the bone marrow and the peripheral blood, which goes along with a suppression of normal hematopoiesis including granulopoiesis, erythropoiesis and thrombocytopoiesis. The prognosis is largely determined by cytogenetic and molecular risk factors, age, performance status and antecedent Myelodysplastic Syndrome (MDS).

With the exception of old and frail patients, most AML patients are eligible for intensive chemotherapy, which is given in curative intent consisting of induction and consolidation therapy. However, despite intensive therapy, the long-term outcome of AML patients remains poor, with less than 30% of patients achieving long lasting remission and even cure. This poor outcome is largely due to refractoriness to induction chemotherapy as well as relapses during and after completion of intensive induction and consolidation therapy. Regarding refractoriness, about 20-30% of AML patients under the age of 60 years and about 50% of older patients fail to attain complete remission (CR) following cytarabine plus anthracycline based standard induction therapy. Regarding relapses, even patients having achieved complete remission are at a high risk of relapse, particularly within the first two years after completion of chemotherapy.

In patients with blast persistence after induction therapy or relapse, allogeneic hematopoietic cell transplantation (allo-HCT) is currently the only treatment strategy to offer the prospect of cure. Outcome of allo-HCT is heavily influenced by the remission state before allo-HCT. With the aim to induce a complete remission (CR) before allo-HCT, salvage chemotherapy regimens are administered in refractory/relapsed patients. Typically, these salvage regimens are based on high dose cytarabine (HiDAC), which is frequently combined with either mitoxantrone (HAM regimen) or fludarabine plus idarubicin (idaFLA regimen). Currently, there is no commonly accepted standard salvage regime, but a large individual patient data meta-analysis and single arm phase-II studies suggest that combination chemotherapy including HiDAC and gemtuzumab ozogamicin, an antibody drug conjugate, are very effective. Since patients with refractory or relapsed AML are candidates for allo-HCT, the main purpose of the salvage regimen is to bridge patients to allo-HCT with induction of a CR before allo-HCT. Therapy resistance in cancer is still poorly understood. Beyond genetic aberrations epigenetic mechanisms are important components of resistance to cancer therapy. Recently, the investigators discovered an epigenetic therapy resistance mechanism in AML (Figure 1). This mechanism might be relevant in up to 50% of relapsed/refractory AML patients. This epigenetic mediated resistance can be successfully overcome in in vitro models by proteasome inhibition. Currently, relapsed and refractory r/r-AML still carries a dismal prognosis. In this multicentre, phase II trial the investigators will analyze efficacy of a novel therapy regimen for r/r-AML.

As detailed above, combination-chemotherapy including GO and HiDAC based chemotherapy is an effective regimen in r/r-AML.

Proteasome inhibitors can restore EZH2 protein levels in vitro and in vivo. The restoration of EZH2 significantly improved efficacy of anti-leukemic therapy. Based on the data mentioned above we combine the treatment efficacy of GO plus cytarabine based chemotherapy with the proteasome inhibitor bortezomib in the B-GA regimen. With such an approach the investigators believe that they can substantially improve treatment results in r/r-AML. Part of the study is a pre-specified biomarker analysis for EZH2 restoration after bortezomib exposure in vitro and in vivo. Accordingly, we will be able to determine whether EZH2 restoration after bortezomib exposure is associated with response and outcome. There have been rare reports of acute diffuse infiltrative pulmonary disease of unknown etiology such as pneumonitis, interstitial pneumonia, lung infiltration and Acute Respiratory Distress Syndrome (ARDS) in patients receiving bortezomib. In particular, 2 patients with r/r-AML given high-dose cytarabine (2 g/m²/day) by continuous infusion in combination with daunorubicin and bortezomib died of ARDS early in the course of therapy. However, in several trials evaluating the combination of bortezomib with standard and high-dose cytarabine in AML patients no toxicity signal was detected, especially with respect to ARDS.

Taken together, the rationale for this trial is based on the high unmet clinical need and strong in vitro evidence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of AML according to WHO-2016 [27] (except acute promyelocytic leukemia) either de novo AML, AML after preceding myelodysplastic or myeloproliferative syndrome (MDS/MPD), and therapy related AML (t-AML) after previous cytotoxic therapy or radiation are eligible either refractory (A) to first line chemotherapy or in first relapse (B), also after stem cell transplantation. FLT3-ITD status, cytogenetics (refractory and relapsed patients), in addition status of core-binding-factor as well as double mutant CEBPA in relapsed patients must be available.

A) Refractory to induction therapy is defined as no CR, CRi (according to standard criteria) [4] after 2 intensive induction cycles of at least 7 days of cytarabine 100-200 mg/m² continuously or an equivalent regimen with cytarabine with total dose not less than 700 mg/m² per cycle and 3 days of an anthracycline/ anthraquinone (e.g. daunorubicin, idarubicin).

B) Relapsed after first line therapy is defined as relapsed AML after CR or CRi (according to standard criteria) after at least one intensive induction and consolidation (including intensive chemotherapy and/or hematopoietic cell transplantation) therapy.

* ECOG performance status ≤ 2
* Discontinuation of prior AML treatment before the start of study treatment (except hydroxyurea or other treatment to control hyperleukocytosis) for at least 10 days for cytotoxic agents and 5 half-lives for non-cytotoxic/ investigational drug treatment preceding the first dose of trial medications
* Age ≥ 18 years
* Pregnancy and childbearing potential:

  * Non-pregnant and non-nursing women of childbearing potential must have a negative serum or urine ß-HCG pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months).
  * Female patients of reproductive age must agree to avoid getting pregnant while on therapy.
  * Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin highly effective methods of birth control during study and for at least 7 months after end of treatment.
  * Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy and must agree to avoid to father a child during study and until 6 months after end of study/treatment.
* Willingness of patient to adhere to protocol specific requirements and capacity to give written informed consent
* Ability of patient to understand the character and individual consequences of clinical Trial
* Following receipt of verbal and written information about the study, the patient must provide signed informed consent before any study related activity is carried out

Exclusion Criteria:

* Acute promyelocytic leukemia (AML M3)
* Acute myeloid leukemia previously treated with gemtuzumab ozogamicin
* Hyperleukocytosis (leukocytes > 30,000/μl) at the time of study entry. These patients should be treated with hydroxyurea and / or receive leukocytapheresis treatment according to routine practice and are only allowed to enter into the study when leukocyte counts of 30,000/μl or below are reached. If hydroxyurea is not sufficient to control hyperleukocytosis i.v. application of 100 mg cytarabine continuously over 24 hours may be discussed with the coordinating investigator or the scientific coordinator
* Known central nervous system manifestation of AML
* uncontrolled or significant cardiovascular disease, including any of the following:

  * History of heart failure NYHA class 3 or 4
  * Left ventricular ejection fraction (LVEF) ≤ 40% by echocardiogram
  * History of uncontrolled angina pectoris or myocardial infarction within 12 months prior to screening
  * History of second (Mobitz II) or third degree heart block or any cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Pregnant or nursing woman
* Chronically impaired renal function (creatinine clearance < 30 ml / min)
* Inadequate liver function (ALT and AST ≥ 2 x ULN), total bilirubin ≥ 1.5 x ULN
* Known liver cirrhosis or history of veno-occlusive disease (VOD)
* HIV infection and/or active hepatitis B or C infection (active hepatitis B defined by HBs Ag positivity, active hepatitis C defined by positive virus load)
* Evidence or history of severe non-leukemia associated bleeding diathesis or coagulopathy
* Uncontrolled active infection
* Concurrent malignancies other than AML with an estimated life expectancy of less than two years
* Known hypersensitivity to cytarabine (AraC) (not including drug fever, conjunctivitis or exanthema)
* Known hypersensitivity to bortezomib, boron or mannitol
* Isolated extramedullary manifestation of AML
* Patients within 100 days after allogeneic stem cell transplantation at the time of Screening
* Patients with clinically relevant Graft-versus-Host-Disease (GvHD) requiring initiation of treatment or treatment escalation within 21 days prior to Screening
* Patients with pre-existing severe neuropathy
* Acute diffuse infiltrative pulmonary disease
* Pericardial disease
* Expected incompliance of patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
CR/CRi rate | two years
  Primary endpoint is the CR/CRi rate (response rate), defined as the proportion of patients achieving a complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) according to ELN 2017 criteria after B-GA treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Müller-Tidow, Prof., MD, Principal Investigator — Medical Director of Internal Medicine V, University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Internal Medicine V, Heidelberg, Baden-Wurttemberg, Germany